CLINICAL TRIAL: NCT06773871
Title: Feasibility and Safety of Exercise in Patients With Low-risk (or Early-stage) Myeloid Cancers and Precursor Conditions (HemEx): a Randomized Controlled Pilot Trial
Brief Title: Feasibility and Safety of Exercise in Patients With Low-risk Myeloid Cancers and Precursor Conditions
Acronym: HemEx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kirsten Grønbæk, Professor, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-23022425
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Myelodysplastic Syndrome; Cytopenia
MeSH Terms: conditions — Myelodysplastic Syndromes; Cytopenia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Usual care
  Interventions: Other: Control
- Exercise intervention (Experimental): High-intensity interval exercise (180 min/week)

INTERVENTIONS:
Other: Exercise — Weekly supervised exercise for 12 weeks followed by 12 weeks of non-supervised exercise
Other: Control — Remain usual activity level
  Arms: Control

SUMMARY:
Somatic mutations as seen in myeloid malignancies can also be detected in healthy, elderly individuals (clonal hematopoiesis of indeterminate potential, CHIP), in patients with unex-plained cytopenia, that do not fulfill the criteria for myeloid malignancy (clonal cytopenia of un-determined significance, CCUS) It has been shown that these conditions predispose to hema-tological cancer. For patients with CCUS, it has been reported that in a 5-year period up to 50-90 % of the patients will progress to myelodysplastic syndrome (MDS) or acute myeloid leu-kemia (AML), both devastating diseases with poor outcomes, especially for the elderly popula-tion. There is currently no treatment available for patients with CCUS besides supporting agents. Since the somatic mutations can be detected up to 10 years before a diagnosis of MDS, it opens the potential for early intervention.

Physical inactivity is associated with multiple solid cancers, and it has been suggested that exercise can prevent for example certain colon- or breast cancers. Studies in mice have shown that exercise can reduce tumor size and incidence of solid cancers, and different mechanisms have been suggested including increased immune cell infiltration, reduced systemic inflamma-tion, and metabolic changes. The mechanisms of disease progression of pre-leukemia and MDS are complex and probably multifactorial, but recent studies suggest that components such as natural killer cells, adipocytes, and inflammatory substances in the bone marrow mi-croenvironment play a crucial role; factors that exercise may modulate. In addition, recent stud-ies have shown that increased bone marrow adipose tissue (BMAT) may create a microenvi-ronment that supports the expansion of leukemic cells and thus may facilitate disease progres-sion, and earlier studies among healthy, younger individuals have shown that exercise can reduce the amount of BMAT significantly.

Therefore, the investigators hypothesize that exercise may prevent or delay the progression from pre-leukemia to leukemia by altering the microenvironment in the bone marrow.

The purpose with this clinical, pilot trial where patients with the preleukemic condition CCUS or early stage of leukemia (i.e., lower-risk MDS) will undergo an individualized exercise interven-tion, is to investigate:

1. whether an exercise intervention and the trial set-up, are feasible and safe in this cohort,
2. potential mechanisms in leukemogenesis affected by exercise in controlling dis-ease progression,
3. and the effect hereof on quality of life and activities of daily living. The above will inform the decision-making on designing a larger randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of either Lower-risk of Myelodysplastic Syndrome or Clonal Cytopenia of undetermined significance(WHO 2022 Classification)
* Written informed consent prior to study procedures
* Performance status ≤ 2
* Age > 18 years old

Exclusion Criteria:

* Physically not able to undergo exercise intervention (e.g., arthrosis, physical disabilities)
* Exercising on a regular basis (i.e., participants must score in the category "low" when screening with International Physical Activity Questionnaire-Short Form; IPAQ-SF27)
* Unwillingness to undergo exercise intervention
* Use of metformin
* Treatment with chemotherapy, therapeutic radiation, or immunosuppressive therapy within the last year
* Treatment with hypomethylating agents
* Any absolute contraindication to undergo cardiopulmonary exercise testing according to working papers from American Heart Association and Danish Society of Cardiology
* Hemoglobin levels < 5.5 mmol OR <6.5 mmol and simultaneous cardiac insufficiency OR pacemaker.
* Blood transfusion-dependent ≥ 8 units of red blood cell transfusion in 16 weeks (IWG 2018-criteria)
* Uncontrolled co-morbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Exercise feasibility: Exercise sessions attendance | From baseline until the end of12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  The number of attended exercise training sessions relative to the number of planned exercise sessions
Exercise feasibility: Recruitment, refusal, and retention rates | From baseline until end of intervention (24 weeks)
  The number of patients recruited to the study, the number of patients who refused to be enrolled in the study, the number of participants that completed the study
Incidence of Adverse Events (AEs) | From baseline until the end of intervention (24 weeks)
  AE will be recorded during trial assessment visits and through medical records. This procedure will concern any AE during the trial period. We will collect patients' self-report of AEs for each trial visit and telephone interview, which may have occurred since the last trial visit and telephone interview.
Incidence of Serious Adverse Events (SAEs) | From baseline until the end of intervention (24 weeks)
  SAE will be recorded during trial assessment visits and through medical records. This procedure will concern any SAE during the trial period. We will collect patients' self-report of SAEs for each trial visit and telephone interview, which may have occurred since the last trial visit and telephone interview.

SECONDARY OUTCOMES:
Changes in peak oxygen consumption (VO2 peak) | From baseline until the end of12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in VO2peak assessed during an incremental exercise test to volitional exhaustion on a bicycle ergometer
Changes in Aerobic Capacity: Peak power output | From baseline until the end of12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in peak power output assessed during an incremental exercise test to volitional exhaustion on a bicycle ergometer
Changes in Muscle strength: Hand grip strength | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in hand grip strength, assessed using a dynamometer
Changes in Functional performance: Habitual gait speed | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in habitual gait speed
Changes in Functional performance: 30 seconds Sit-to-stand | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in the number of stands from sitting position that can be performed during 30 seconds
Changes in Body composition and anthropometrics: Body mass | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in body mass
Changes in Body composition and anthropometrics: Total lean mass | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in total lean mass assessed by dual energy x-ray absorptiometry (DXA)
Changes in Body composition and anthropometrics: Total fat mass | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in total fat mass assessed by DXA
Changes in Body composition and anthropometrics: Bone mineral density | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in bone mineral density assessed by DXA
Changes in Blood biochemistry: C-reactive protein | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting C-reactive protein levels in blood
Changes in Blood biochemistry: Insulin | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting insulin blood levels
Changes in Blood biochemistry: Glucose | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting glucose blood levels
Changes in Blood biochemistry: Triglycerides | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting triglycerides blood levels
Changes in Blood biochemistry: LDL-Cholesterol | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting LDL-cholesterol blood levels
Changes in Blood biochemistry: HDL-Cholesterol | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting HDL-cholesterol blood levels
Changes in Blood biochemistry: Total Cholesterol | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting Cholesterol blood levels
Changes in Blood biochemistry: HbA1c | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting HbA1c blood levels
Changes in Blood biochemistry: total bilirubin | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting total bilirubin blood levels
Changes in Blood biochemistry: Vitamin D (25-Hydroxy-Vitamin D(D3+D2)) | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting Vitamin D (25-Hydroxy-Vitamin D(D3+D2)) blood levels
Changes in Blood biochemistry: insulin growth factor 1 (IGF-1) | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting insulin growth factor 1 (IGF-1) blood levels
Changes in Blood biochemistry: human growth hormone (HGH) | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting human growth hormone (HGH) blood levels
Changes in Blood biochemistry: sex hormones (estrogen, progesterone and testosterone) | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting human sex hormones (estrogen, progesterone and testosterone)blood levels
Changes in Cytokine levels in blood: Interleukin-6 | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting Interleukin-6 blood levels
Changes in Cytokine levels in blood: Tumor-necrosis-factor alpha (TNFalpha) | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting TNFalpha blood levels
Changes in Patient-reported symptomatic adverse events | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Patient-reported symptomatic adverse events, assessed using the using the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Inflammatory markers in Bone marrow (BM) and peripheral blood | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in the inflammatory markers INF-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, TNF-α, adiponectin and leptin in bone marrow aspirate and peripheral blood
Regulate the immune cell composition in the BM | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in immune cell composition in the BM measured by flow cytometry
Change the variant allele frequency (VAF) | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in VAF detected with targeted next generation sequencing (NGS)
Alter the composition of BMAT | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in BMAT composition
Ifluence on the cytopenia(s) | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in blood cell counts (i.e., hemoglobin, white blood cell count, platelet count, absolute neutrophil count, lymphocyte count, basophil count, eosinophil count, monocyte count, reticulocyte count, peripheral blood blast count, red cell)
Changes in Blood biochemistry: Lactate dehydrogenase (LDH) | From baseline until the end of 12 weeks of supervised exercise. And after 12 weeks of no supervised exercise.
  Changes in resting Lactate dehydrogenase (LDH) blood levels

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen, Denmark
  - Rigshospitalet, Copenhagen